

### Statistical Analysis Plan

NCT Number: NCT04804813

Title: CABOMETYX Tablets General Drug Use Results Surveillance Study "Renal Cell

Carcinoma"

Study Number: Cabozantinib-5001

Document Version and Date: Original version / 20-MAY-2024

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

Note; This document was translated into English as the language on original version was Japanese.

### Statistical Analysis Plan



Akeda Pharmaceutical Con Head of Biostatistics Office

Original: Prepared on May 20, 2024

### TABLE OF CONTENTS

| L | ist of T | Геrm | s and Abbreviations | 3 |
|---|---|---|---|---|
| A | nalysis | s Set | ts | 5 |
| N | umber | of | digits to be displayed | 6 |
| S | afety s | peci | fication (Important identified risks, important potential risks, and important missing | |
| | info | rmat | ion) | 7 |
| 1 | Num | ıber | of medical institutions surveyed, number of patients enrolled, and patient composition | 8 |
| | | | position of patients | ز<br>8 |
| 2 | Patie | ent c | haracteristics | 10 |
| | 2.1 | Pati | lent characteristics | 10 |
| 3 | Deta | ils o | of treatment | 13 |
| | 3.1 | Adr | ministration status of Cabometyx | 13 |
| | 3.2 | Stat | tus of Administration of Therapeutic Drugs for Renal Cell Carcinoma Other than | |
| | | Са | abometyx | 13 |
| | 3.3 | Stat | abometyxtus of Administration of Nivolumabtus of Administration of Nivolumab | 14 |
| | 3.4 | Obs | servation period radiotherapy | 14 |
| 4 | Matt | ters ( | concerning safety | 15 |
| | | | currence Status of Adverse Events and Adverse Drug Reactions/Infections | 15 |
| | 4. | 1.1 | Data on adverse events | 15 |
| | 4.1 | 1.2 | Status of onset of ADRs/infections | 16 |
| | 4.1 | 1.3 | Occurrence Status of Adverse Events and Adverse Drug Reactions/Infections Included in | |
| | | | Safety Specifications | 17 |
| | 4.2 | Inci | idences of adverse events and adverse drug reactions/infections in patients excluded from | |
| | | sa | fety evaluation | 19 |
| | 4.2 | 2.1 | Incidences of adverse events in patients excluded from safety evaluation | 19 |
| | 4.2 | 2.2 | Occurrence of ADRs/infections in patients excluded from safety evaluation | 19 |
| | 4.3 | Stat | tus of adverse events and onset of adverse reactions/infections by seriousness, CTCAE | |
| | | Gı | rade (worst value), timing of onset, outcome, and causal relationship with Cabometyx | 19 |
| | 4 | 3.1 | Occurrence status of adverse events by seriousness, CTCAE Grade (worst value), time to | |
| 9 | 2/- | | onset, outcome, and causal relationship to Cabometyx | 19 |
| | 4.3 | 3.2 | Occurrence status of ADRs/infections by seriousness, CTCAE Grade (worst value), time | |
| | | | to onset, and outcome | 21 |
| | 4.3 | 3.3 | Status of occurrence of adverse events and adverse reactions/infections specified in the | |
| | | | safety specification by seriousness, CTCAE Grade (worst value), time to onset, outcome, | |
| | | | and causal relationship with Cabometyx | 22 |

| 4.3.4 S | Status of occurrence of adverse events and adverse reactions/infections by CTCAE | |
|---|---|---|
| ( | Grade (worst value) and by administration status of Cabometyx | 23 |
| 4.3.5 | Time to initial onset of adverse events and adverse drug reactions/infections included | in 26 ons 26 26 |
| ť | he safety specifications | 26 |
| 4.4 Status | s of administration of Cabometyx due to adverse events and adverse reactions/infection | ons 26 |
| 4.4.1 A | Administration status of Cabometyx due to adverse events | 26 |
| 4.4.2 A | Administration status of Cabometyx due to adverse reactions/infections | 26 |
| 4.4.3 A | Administration status of Cabometyx due to adverse events and adverse | \@ ` |
| r | eactions/infections specified in the safety specifications | 27 |
| 4.5 Factor | Administration status of Cabometyx due to adverse events and adverse eactions/infections specified in the safety specifications | 28 |
| 4.5.1 | Status of occurrence of adverse events and adverse drug reactions/infections by patien | nt |
| ł | packground and treatment characteristics | 28 |
| 4.5.2 I | ncidences of ADRs/infections by gender | 31 |
| 4.5.3 I | ncidences of ADRs and infections by age group | 31 |
| | Status of occurrence of ADRs/infections by presence/absence of hepatic impairment | |
| | Status of occurrence of ADRs/infections by presence/absence of renal impairment | |
| 5 Matters co | ncerning efficacyumor effect | 33 |
| 5.1 Antitu | umor effect | 33 |
| 5.2 Tumo | r response by patient background factors and treatment factors | 33 |
| 6 Incidences | of adverse reactions/infections in the additional pharmacovigilance plan | 36 |
| | ences of adverse reactions and infections in the additional pharmacovigilance plan | |
| (Atta | ached Form 12) | 36 |
| 7 Incidence | of adverse reactions/infections in post-marketing surveillance, etc. | 37 |
| 7.1 Incide | ence of adverse reactions/infections in post-marketing surveillance, etc. (Attached For | rm |
| 15). | | 37 |
| 8 Case summ | nary in post-marketing surveillance, etc | 39 |
| 8.1 Case : | summaries from post-marketing surveillance, etc. (Attached Form 16) | 39 |
| - v | story (version control) | 40 |
| [Amandir 1] | Comparison Table of Changes | 1 |
| 15)<br>8 Case sumn<br>8.1 Case s<br>Preparation hi | nary in post-marketing surveillance, etcsummaries from post-marketing surveillance, etc. (Attached Form 16) | 37<br>39<br>39 |

### **List of Terms and Abbreviations**

- This drug: CABOMETYX Tablets is abbreviated as this drug.
- Adverse event: AE that occurred after receiving Cabometyx.
- Adverse reactions, etc.: Acronym of the term "adverse reactions/infections." Adverse events for
  which the causal relationship with Cabometyx is other than "Not related" in the assessment of the
  investigator. In this statistical analysis plan, the term "adverse drug reactions/infections" is used in
  the title, and "adverse drug reactions, etc." is used in the text and tables.
- Serious adverse events: Adverse events assessed as "serious" by the investigator. Events listed in the MedDRA code list (PT code) of the Important Medical Events List will be handled as serious even if the investigator's assessment is "non-serious."
- Related to Cabometyx: AEs other than 'Not Related' for Cabometyx will be handled as 'Related' and AEs assessed as 'Not Related' for Cabometyx will be handled as 'Not Related'.
- Summary statistics: A general term for the number of subjects, mean, standard deviation, maximum, minimum, and quartiles.
- Patients whose CRFs were not collected: Registered patients whose CRFs were not collected.
- Patients whose CRFs were collected: Registered patients whose CRFs were collected.
- Days after treatment: Day -1 is defined as the day before the first dose of Cabometyx, and Day 1 is defined as the day of the first dose of Cabometyx.
- Duration of Cabometyx treatment (days): Calculated as the end date of Cabometyx treatment start date of Cabometyx treatment +1. However, if "Continuing after the end of the observation period" is selected for the administration status of Cabometyx, the date of last observation will be calculated as the end date of administration of Cabometyx.
- Timing of onset of adverse events (or adverse reactions, etc.): Calculated as the date of onset of adverse events (or adverse reactions, etc.) the start date of the first administration of Cabometyx
- Cabometyx monotherapy patients: patients who received only Cabometyx without concomitant use
  of nivolumab.
- Patients receiving nivolumab combination therapy: Patients receiving Cabometyx in combination with nivolumab.
- Duration of disease:

- Actual number (unit: year) = (Year of the first administration of Cabometyx Year of the diagnosis of renal cell carcinoma) + (Month of the first administration of Cabometyx - Month of the diagnosis of renal cell carcinoma)/12 (Rounded off to one decimal place). If the month of diagnosis is unknown, it should be calculated as January of the year described. If the year of diagnosis is unknown, the data will be considered missing.
- BMI (kg/m<sup>2</sup>): Calculated with weight (kg)/height (m)<sup>2</sup> (rounded to one decimal place).
- Patients with hepatic impairment: Patients with complication specified as MedDRA SMQ "liver disorder (narrow)" in the column of disease name
- Renal Impairment: patients with complication specified as Takeda MedDRA query (TMQ) (Renal Disease) in the disease torre (\*\* 11 Disease) in the disease term field
- RDI (Relative Dose Intensity): Calculated using the following formula.
- RDI (%) = (Total dose of Cabometyx (mg)/Total duration of treatment (days))/ $60 \times 100$ However, for patients treated with nivolumab combination therapy, the calculation is performed Property of Takeda. For non-commercial use only using the following formula.

RDI (%) = (Total dose of Cabometyx (mg)/Total duration of treatment (days))/40  $\times$ 100

### **Analysis Sets**

In this study, the "safety analysis set" and "effectiveness analysis set" will be established as analysis

evaluable for the safety." Patients with locked CRFs who meet the following conditions will be excluded from the safety analysis set.

• Cabometyx naïve
• Administration before again and and an analysis of the ana

- Enrollment outside the enrollment period
- Enrollment after the start date of prescription of Cabometyx (31 days)
- · Onset status of adverse event unknown
- · Withdrew consent
- Effectiveness analysis set

Defined as "Patients evaluable for effectiveness without major protocol deviation among patients eligible for safety evaluation." Patients eligible for the safety evaluation who meet any of the following conditions

### Number of digits to be displayed

e data.

aree data.

6

### Safety specification (Important identified risks, important potential risks, and important missing information)

- Important identified risks
- icable Terms of Use Hepatic failure, hepatic function disorder: Events falling under MedDRA PT included in any of the following MedDRA SMQs:
  - ·Drug related hepatic disorders severe events only (narrow)
  - ·Cholestasis and jaundice of hepatic origin (narrow)
  - ·LIVER LABORATORY TESTS, SIGNS AND SYMPTOMS (NARROW)
  - Pancreatitis: Events that fall under MedDRA PT included in MedDRA SMQ "acute pancreatitis (narrow)" or any of the following MedDRA PTs:
- ed, Lip all, Pancreat all guides only and guides on guid ·Amylase increased, Amylase abnormal, Lipase increased, Lipase abnormal, Pancreatic enzymes increased, Pancreatic enzyme test abnormal, Pancreatic enzyme abnormality,

### 1 Number of medical institutions surveyed, number of patients enrolled, and patient composition

### 1.1 Disposition of patients

Analyzed: All registered patients (registered patients)

Analysis item: Enrolled patients

Study site

Patients with no CRF collected

CRF collected patients

Patients excluded from safety evaluation \*

Reason for exclusion (multiple counts) [ No administration, administration

before the contract period,

enrollment outside the enrollment period, enrollment after 31 days from the start date of prescription of Cabonetyx, occurrence of adverse

events unknown, consent

withdrawal]

Safety analysis set

Patients excluded from efficacy evaluation

Reason for exclusion

[Other than target disease, deveation of

exclusion criteria]

Effectiveness analysis set

Analytical

method:

Property of Lakeda. For

For the above analytical variables, the following analyses will be performed, and a diagram of patient composition will be prepared.

The number of study sites will also be shown for patients enrolled. A medical institution with different clinical departments in the study will be counted as one medical institution.

If there is no patient meeting the reason for exclusion, 0 patient will be displayed. For patients excluded from the safety evaluation and efficacy evaluation, the number of patients by reason for exclusion will be tabulated and a list will be prepared.

\*"Patients excluded from safety evaluation" refer to patients excluded from "patients included in safety evaluation" among patients whose case study forms are collected. Similarly, "patients excluded from efficacy evaluation" refer to patients who are excluded from the" efficacy evaluation population" among the "safety evaluation population."

(1) Calculation of frequencies

Propary of Lakeda: For non-commercial use only and subject to the applicable Terms of use

#### 2 **Patient characteristics**

#### 2.1 **Patient characteristics**

Analyzed: Safety analysis set

Analysis item: Sex

-oo, 85<= - <=Max]

[Min<= - <15, 15<= - <65, 65<= - <75, 75<= - <85, 85<= - <=Max]

[Min<= - <1, 1<= - <=Max]

[Min<= - <1, 1<= - <=Max]

Clear cell Age (years)

Duration of disease (years)

[Clear cell, non-clear cell, unknown] Histological diagnosis

[I, II, III, IV, unknown] Clinical Stage

(At the start of administration)

[Outpatient, Inpatient] Treatment category

(At the start of administration)

Karnofsky Performance Status

Scale (at the start of treatment)

[favorable, intermediate, poor, unknown] IMDC Risk Categorization

(At the start of administration)

Metastasis [Absent, present, unknown]

(At the start of administration)

Destination of metastasis [Brain, lung, liver, bone, lymph node, others]

(multiple counts)

Height (cm) [Min<= - <140, 140<= - <150, 150<= - <160,

160<= - <170, 170<= - <= Max, not measured]

[Min<= - <50, 50<= - <65, 65<= - <=Max, not

measured]

[Min<= - <18.5, 18.5<= - <25.0, 25.0<= -

<30.0, 30.0 <= - <= Max

[Absent, present]

History of radiotherapy prior to

ght (en Weight (kg) BMI(kg) the start of Cabometyx

Anatomical Location (Count

[Brain, lung, liver, bone, lymph node, others]

Presence/absence of prior [Absent, present] systemic drug therapy for renal [Sunitinib, pazopanib, sorafenib, temsirolimus, elimbolimus, axitinib, interferon alpha, nivolumab, ipilimumab + r<sup>2</sup> pembrolimus cell carcinoma before the start of Cabometyx (not including preoperative or postoperative adjuvant drug therapy) History of systemic drug therapy for renal cell carcinoma before the start of Cabometyx (multiple pembrolizumab, avelumab + axitinib, others] counts) Treatment or surgery for renal cell [Absent, present] carcinoma prior to the start of Cabometyx [Total nephrectomy, partial nephrectomy, no Nephrectomy nephrectomy] The status of treatment or surgery for renal cell carcinoma before the start of Cabometyx administration is "Present." Presence/absence of history of [Absent, present] preoperative or postoperative adjuvant drug therapy before the start of administration of Cabometyx When nephrectomy (yes/no) is "total nephrectomy" or "partial nephrectomy" History of preoperative or [Preoperative and postoperative] postoperative adjuvant drug therapy before the start of administration of Cabometyx (duplicate counting) Presence or absence of medical [Absent, present] history Presence or absence of [Absent, present] complications Presence or absence of hepatic [Absent, present]

impairment

Property of Lakedai. For

Presence or absence of renal [Absent, present]

Property of Takeda. For non-commercial use only and subject to the applicable Temes of use

12

#### **Details of treatment** 3

#### 3.1 Administration status of Cabometyx

Analyzed: Safety analysis set

icable reims of Use Analysis item: Cabometyx Starting Dose (mg) [60 mg/day, 40 mg/day, 20 mg/day, 20

mg/day every other day, others]

Duration of treatment (days)

Cabometyx Mean dose (mg/day)

RDI(%)

Presence or absence of dose reduction [Absent, present]

Dose after dose reduction (multiple

counts) [40 mg/day, 20 mg/day, others]

Cabometyx Monotherapy Cases [20 mg/day, 20 mg/day every other day,

Patients receiving combination

therapy with nivolumab

Presence or absence of interruption [Absent, present] [Absent, present] Discontinuation of Cabometyx

Reason for discontinuation (multiple

counts)

[Treatment goal achieved, adverse event onset, transfer to another hospital, etc., the

patient no longer visits the hospital,

pregnancy, lack of efficacy (including PD),

other]

Analytical

method:

For the above analytical variables, frequency tabulation of categorical data and summary statistics of continuous data will be calculated. This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

### Status of Administration of Therapeutic Drugs for Renal Cell Carcinoma Other than Cabometyx

Analyzed: Safety analysis set

Analysis item: Presence/absence of concomitant drugs [Absent, present]

for the primary disease administered

during the observation period Drug name (duplicate counting)

Analytical For the above analytical variables, frequency tabulations of categorical data will be

method: calculated. This tabulation will be performed for the overall population and by

patients receiving Cabometyx monotherapy and patients receiving nivolumab

combination therapy.

#### 3.3 Status of Administration of Nivolumab

applicable Terms of Use Patients receiving combination therapy with nivolumab among patients included in Analyzed:

safety evaluation

Duration of nivolumab treatment (days) Analysis item:

For the above analytical variables, summary statistics of continuous data will be Analytical

method: calculated.

### 3.4 Observation period radiotherapy

Analyzed: Safety analysis set

Analysis item: Presence/absence of radiotherapy [Absent, present]

during the observation period

[Brain, lung, liver, bone, lymph node, Anatomical Location (Count Multiple)

For the above analytical variables, frequency tabulations of categorical data will be Analytical

performant and performance of the state of t calculated. This tabulation will be performed for the overall population and by method:

patients receiving Cabometyx monotherapy and patients receiving nivolumab

### **Matters concerning safety**

#### 4.1 Occurrence Status of Adverse Events and Adverse Drug Reactions/Infections

### 4.1.1 Data on adverse events

Analytical method:

Analyzed: Safety analysis set

Analysis item: Adverse Events

> For the above analytical variable, the following analyses should be performed. This tabulation will be performed for the overall population and by patients to the applicat receiving Cabometyx monotherapy and patients receiving nivolumabcombination therapy.

- (1) Number of subjects with adverse events
- (2) Number of adverse events
- (3) Incidence of adverse events
- (4) Type of Adverse Event

The following accounting methods will be used for each analysis.

[Number of patients with adverse events]

Number of patients with AEs.

[Number of adverse events]

Number of adverse events experienced. When the same adverse event occurred more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

It is calculated as the number of patients with adverse events/the number of patients evaluated for safety ×100.

[Type of adverse event]

- Adverse events will be coded using the MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
- Property of Takedai. For non-c For SOC, the number of patients with adverse events and the incidence of adverse events should be described in SOC internationally agreed order. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC.
  - For PT, the number of patients with adverse events and the incidence will be described in ascending order of PT code. If the same PT occurs more than once in the same subject, the subject will be counted as 1 subject in the PT.

### 4.1.2 Status of onset of ADRs/infections

Analyzed: Safety analysis set

Analysis item: Adverse Reactions, etc.

Analytical method: For the above analytical variable, the following analyses should be performed.

Applicable Terms of Use This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

(1) Number of patients with adverse drug reactions, etc.

- (2) Number of adverse drug reactions
- (3) Incidence of adverse drug reactions, etc.
- (4) Type of adverse drug reaction, etc.

The following accounting methods will be used for each analysis.

[Number of patients with adverse drug reactions, etc.]

Number of patients with adverse drug reactions, etc.

[Number of adverse drug reactions]

Number of adverse drug reactions, etc. that occurred. When the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse drug reactions, etc.]

Calculate with the number of patients with adverse reactions, etc./the number of patients evaluated for safety ×100.

[Types of adverse drug reactions, etc.]

- Adverse drug reactions will be coded using MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
- For SOC, the number of patients with adverse drug reactions, etc. and the incidence should be described in the order of SOC international consensus. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC.
- Property of Takedai. For non-comi For PT, the number of patients with adverse drug reactions, etc. and the incidence should be entered in ascending order of PT code. If the same PT occurs more than once in the same subject, the subject will be counted as 1 subject in the PT.

### 4.1.3 Occurrence Status of Adverse Events and Adverse Drug Reactions/Infections Included in **Safety Specifications**

### 4.1.3.1 Incidences of adverse events included in safety specifications (tabulation by risk)

Analyzed: Safety analysis set

Analysis item: Adverse events included in the important identified risks (Hepatic failure,

hepatic function disorder, pancreatitis) in the safety specifications

Stratification items: Total

> Seriousness [Serious, non-serious]

For the above analytical variables, the following analyses should be Analytical method:

> performed for each risk and each of the subgroups of the stratification factors. The risks to be covered shall be in accordance with the definitions described in the safety specifications (important identified risks). This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

[Number of patients with adverse events]

Number of patients with AEs.

[Number of adverse events]

Number of adverse events experienced. When the same adverse event occurred more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

It is calculated as the number of patients with adverse events/the number of patients evaluated for safety ×100.

[Type of adverse event]

- Adverse events will be coded using the MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
- Property of Takedai. For non-c' For SOC, the number of patients with adverse events and the incidence of adverse events should be described in SOC internationally agreed order. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC. However, if different in each stratification category, the subject will be counted as 1 subject in each category. For the last stratification item, one item will be adopted in accordance with the order of priority.
  - For PT, the number of patients with adverse events and the incidence will be described in ascending order of PT code. If the same PT occurs

more than once in the same subject, the subject will be counted as 1 subject in the PT. However, if different in each stratification category, the Terms of Use subject will be counted as 1 subject in each category. For the following stratification items, 1 case will be adopted in accordance with the order of priority.

Seriousness: Serious → Non-serious

### Incidences of ADRs/infections included in safety specifications (tabulation by risk) 4.1.3.2

Analyzed: Safety analysis set

Analysis item: Adverse reactions, etc. corresponding to important identified risks (Hepatic

failure, hepatic function disorder, pancreatitis) in safety specifications

Stratification items: Total

Property of Lakedai. For hon

[Serious, non-serious] Seriousness

Analytical method: For the above analytical variables, the following analyses should be

> performed for each risk and each of the subgroups of the stratification factors. The risks to be covered shall be in accordance with the definitions described in the safety specifications (important identified risks). This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

[Number of patients with ADRs]

Number of patients with adverse drug reactions, etc.

[Number of adverse drug reactions]

Number of adverse drug reactions, etc. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

[Incidence of ADRs]

Calculate with the number of patients with adverse reactions, etc./the number of patients evaluated for safety ×100.

[Type of adverse drug reaction, etc.]

- Adverse drug reactions will be coded using MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
- For SOC, the number of patients with adverse drug reactions, etc. and the incidence should be described in the order of SOC international consensus. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC. However, if different in each

stratification category, the subject will be counted as 1 subject in each category. For the last stratification item, one item will be adopted in accordance with the order of priority.

For PT, the number of patients with adverse drug reactions, etc. and the
incidence should be entered in ascending order of PT code. If the same
PT occurs more than once in the same subject, the subject will be
counted as 1 subject in the PT. However, if different in each stratification
category, the subject will be counted as 1 subject in each category. For
the following stratification items, 1 case will be adopted in accordance
with the order of priority.

Seriousness: Serious → Non-serious

# 4.2 Incidences of adverse events and adverse drug reactions/infections in patients excluded from safety evaluation

### 4.2.1 Incidences of adverse events in patients excluded from safety evaluation

Analyzed: Patients excluded from safety evaluation

Analysis item: Adverse Events

Analytical method: For the above analytical variable, analyses should be performed in the same

manners as in Section 4.1.1. This tabulation is for all subjects only.

### 4.2.2 Occurrence of ADRs/infections in patients excluded from safety evaluation

Analyzed: Patients excluded from safety evaluation

Analysis item: Adverse Reactions, etc.

Analytical method: For the above analytical variable, analyses should be performed in the same

manners as in Section 4.1.2. This tabulation is for all subjects only.

4.3 Status of adverse events and onset of adverse reactions/infections by seriousness, CTCAE Grade (worst value), timing of onset, outcome, and causal relationship with Cabometyx

4.3.1 Occurrence status of adverse events by seriousness, CTCAE Grade (worst value), time to onset, outcome, and causal relationship to Cabometyx

Analyzed: Safety analysis set

Analysis item: Adverse Events

Stratification items: Total

Seriousness [Serious, non-serious]

CTCAE Grade (worst) [Grade1, Grade2, Grade3, Grade4, Grade5]

[Grade  $\geq$  3]

Time of onset (Day) [1<= - <=21, 22<= - <=84, 85<= - <=168,

 $169 \le - \le Max$ 

cerms of Use [Recovered/resolved, recovering/resolving, Outcome

not recovered/not resolved,

recovered/resolved with sequelae, death

(due to the event), unknown]

Relationship to Cabometyx [Related, Not Related]

Analytical method:

For the above analysis set, the following analyses will be performed in each stratum of the stratification factor. This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

- (1) Number of subjects with adverse events
- (2) Number of adverse events
- (3) Incidence of adverse events
- (4) Type of Adverse Event

The following accounting methods will be used for each analysis.

[Number of patients with adverse events]

Number of patients with AEs.

[Number of adverse events]

Number of adverse events experienced. When the same adverse event occurred more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

It is calculated as the number of patients with adverse events/the number of patients evaluated for safety ×100.

[Type of adverse event]

- Adverse events will be coded using the MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
- Property of Takedai. For non-c', For SOC, the number of patients with adverse events and the incidence of adverse events should be described in SOC internationally agreed order. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC. However, one case of the same SOC will be adopted in accordance with the last priority.
  - In PT, the number of patients with adverse events and the incidence of them will be entered in ascending order of PT code. If the same PT

occurs more than once in the same subject, the subject will be counted as 1 subject in the PT. However, 1 case of the same PT will be adopted in Timing of onset (days): 1-21 days →22 to 84 days →85 to 168 days →20 days

Outcome: Fatal (due to the event) → recovered recovered → reco

CTCAE Grade (worst value):

Grade5→Grade4→Grade3→Grade2→Grade1

Causal relationship with Cabometyx: Related → Not related

### 4.3.2 Occurrence status of ADRs/infections by seriousness, CTCAE Grade (worst value), time to onset, and outcome

Analyzed: Safety analysis set

Analysis item: Adverse Reactions, etc.

Stratification items: Total

> Seriousness [Serious, non-serious]

CTCAE Grade (worst) [Grade1, Grade2, Grade3, Grade4, Grade5]

[Grade  $\geq$  3]

Time of onset (Da [1<= - <=21, 22<= - <=84, 85<= - <=168,

 $169 \le - \le Max$ 

[Recovered/resolved, recovering/resolving,

not recovered/not resolved,

recovered/resolved with sequelae, death

(due to the event), unknown]

Property of Lakeda.

Outcome

Analytical method: For the above analysis set, the following analyses will be performed in each stratum of the stratification factor. This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

- (1) Number of patients with adverse drug reactions, etc.
- (2) Number of adverse drug reactions
- (3) Incidence of adverse drug reactions, etc.
- (4) Type of adverse drug reaction, etc.

The following accounting methods will be used for each analysis.

[Number of patients with ADRs]

Number of patients with adverse drug reactions, etc.

### [Number of adverse drug reactions]

 Number of adverse drug reactions, etc. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

### [Incidence of ADRs]

• Calculate with the number of patients with adverse reactions, etc./the number of patients evaluated for safety ×100.

[Type of adverse drug reaction, etc.]

- Adverse drug reactions will be coded using MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
- For SOC, the number of patients with adverse drug reactions, etc. and the incidence should be described in the order of SOC international consensus. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC. However, one case of the same SOC will be adopted in accordance with the last priority.
- In PT, the number of patients with adverse drug reactions, etc. and the incidence thereof should be entered in ascending order of PT code. If the same PT occurs more than once in the same subject, the subject will be counted as 1 subject in the PT. However, 1 case of the same PT will be adopted in the following order of priority.

Seriousness: Serious → Non-serious

CTCAE Grade (worst value):

Grade5→Grade4→Grade3→Grade2→Grade1

Timing of onset (days): 1-21 days  $\rightarrow$ 22 to 84 days  $\rightarrow$ 85 to 168 days  $\rightarrow$   $\geq$  169 days

Outcome: Fatal (due to the event)  $\rightarrow$  recovered with sequelae  $\rightarrow$  not recovered  $\rightarrow$  recovering  $\rightarrow$  recovered  $\rightarrow$  unknown

- 3.3 Status of occurrence of adverse events and adverse reactions/infections specified in the safety specification by seriousness, CTCAE Grade (worst value), time to onset, outcome, and causal relationship with Cabometyx
- 4.3.3.1 Occurrence status of adverse events specified in the safety specification by seriousness, CTCAE Grade (worst value), time to onset, outcome, and causal relationship to Cabometyx

Analyzed:

Safety analysis set

Analysis item: Adverse events included in the important identified risks (Hepatic failure,

hepatic function disorder, pancreatitis) in the safety specifications

Analytical method: For the above analytical variable, analyses should be performed in the same

manners as in Section 4.3.1.

# 4.3.3.2 Occurrence status of ADRs/infections specified in safety specifications by seriousness, CTCAE Grade (worst value), time to onset, and outcome

Analyzed: Safety analysis set

Analysis item: Adverse reactions, etc. corresponding to important identified risks (Hepatic

failure, hepatic function disorder, pancreatitis) in safety specifications

Analytical method: For the above analytical variable, analyses should be performed in the same

manners as in Section 4.3.2.

# 4.3.4 Status of occurrence of adverse events and adverse reactions/infections by CTCAE Grade (worst value) and by administration status of Cabometyx

### 4.3.4.1 Occurrence status of adverse events by CTCAE Grade (worst value) and Cabometyx administration status

Analyzed: Safety analysis set

Analysis item: AEs with (Discontinuation (except interruption), interruption, dose reduction)

if Cabometyxdose changed

Stratification items: Total

Property of Takedai. For not

CTCAE Grade (worst) [Grade1, Grade2, Grade3, Grade4, Grade5]

[Grade  $\geq$  3]

Analytical method: For the above analysis set, the following analyses should be performed by

stratum of the stratification factor and by administration status of Cabometyx (Discontinuation (except interruption), interruption, dose reduction). This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab

combination therapy.

(1) Number of subjects with adverse events

(2) Number of adverse events

(3) Incidence of adverse events

(4) Type of Adverse Event

The following accounting methods will be used for each analysis.

[Number of patients with adverse events]

• Number of patients with AEs.

[Number of adverse events]

 Number of adverse events experienced. When the same adverse event occurred more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse events]

 It is calculated as the number of patients with adverse events/the number of patients evaluated for safety ×100.

[Type of adverse event]

- Adverse events will be coded using the MedDRA/J. Data will be broadly
  classified by SOC, and tabulated by PT within the SOC. If the SOC is
  "investigations," they will be summarized by HLGT (Sort in ascending
  order of HLGT code, but not output) and by PT.
- For SOC, the number of patients with adverse events and the incidence of adverse events should be described in SOC internationally agreed order. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC. However, one case of the same SOC will be adopted in accordance with the last priority.
- In PT, the number of patients with adverse events and the incidence of them will be entered in ascending order of PT code. If the same PT occurs more than once in the same subject, the subject will be counted as 1 subject in the PT. However, 1 case of the same PT will be adopted in the following order of priority.

CTCAE Grade (worst value):

Grade5→Grade4→Grade3→Grade2→Grade1

# 4.3.4.2 CTCAE Grade (worst value), occurrence status of adverse reactions/infections by administration status of Cabometyx

Analyzed: Safety analysis set

Analysis item: Adverse reactions, etc. of (Discontinuation (except interruption), interruption,

dose reduction) because there was presence or absence of dose change for

Cabometyx

Stratification items: Total

CTCAE Grade (worst) [Grade1, Grade2, Grade3, Grade4, Grade5]

[Grade  $\geq$  3]

Analytical method:

For the above analysis set, the following analyses should be performed by stratum of the stratification factor and by administration status of Cabometyx (Discontinuation (except interruption), interruption, dose reduction). This tabulation will be performed for the overall population and by patients

receiving Cabometyx monotherapy and patients receiving nivolumab icable Terms of Use combination therapy.

- (1) Number of patients with adverse drug reactions, etc.
- (2) Number of adverse drug reactions
- (3) Incidence of adverse drug reactions, etc.
- (4) Types of adverse drug reactions, etc.

The following accounting methods will be used for each analysis.

[Number of patients with adverse reactions, etc.]

Number of patients with adverse drug reactions, etc.

[Number of adverse drug reactions]

Number of adverse drug reactions, etc. If the same adverse drug reaction, etc. occurred multiple times in the same patient, the total number of events will be tabulated.

[Incidence of adverse drug reactions, etc.]

Calculate with the number of patients with adverse reactions, etc./the number of patients evaluated for safety ×100.

[Types of adverse drug reactions, etc.]

- Adverse drug reactions will be coded using MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
- For SOC, the number of patients with adverse drug reactions, etc. and the incidence should be described in the order of SOC international consensus. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC. However, one case of the same SOC will be adopted in accordance with the last priority.
- Property of Takedai. For non-cor For PT, the number of patients with adverse drug reactions, etc. and the incidence should be entered in ascending order of PT code. If the same PT occurs more than once in the same subject, the subject will be counted as 1 subject in the PT. However, 1 case of the same PT will be adopted in the following order of priority.

CTCAE Grade (worst value):

Grade5→Grade4→Grade3→Grade2→Grade1

### 4.3.5 Time to initial onset of adverse events and adverse drug reactions/infections included in the safety specifications

Analyzed: Patients with adverse events or adverse drug reactions included in the safety

specifications among the patients included in the safety evaluation

Analysis item: Time to initial onset of adverse events included in the important identified risk

(Hepatic failure, hepatic function disorder, pancreatitis) in the safety

specifications (days)

Time to initial onset of ADRs, etc. corresponding to the important identified risks (Hepatic failure, hepatic function disorder, pancreatitis) in the safety

specifications (days)

Analytical method: For the above analytical variables, summary statistics will be calculated for

the time of the first onset (Day). This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and

patients receiving nivolumab combination therapy.

### 4.4 Status of administration of Cabometyx due to adverse events and adverse reactions/infections

### 4.4.1 Administration status of Cabometyx due to adverse events

Analyzed: Safety analysis set

Analysis item: Adverse Events

Stratification items: Presence or absence of dose change [Absent, present]

for Cabometyx

Breakdown of changes (duplicate [Discontinued (except for

counting) interruption), interrupted, dose

reduced, unknown]

Analytical method: For the above analysis set, frequencies of the number of adverse events will

be tabulated for each CTCAE Grade (worst value) of adverse events and stratification by the stratification factor. Similar frequency tabulation will be performed for total and CTCAE Grade  $\geq$  3. For the incidence of events by

stratification factor, the denominator will be the number of events by CTCAE Grade (worst value). This tabulation will be performed for the overall

population and patients treated with Cabometyx monotherapy and patients

treated with nivolumab combination therapy separately.

### 4.4.2 Administration status of Cabometyx due to adverse reactions/infections

Analyzed: Safety analysis set

Analysis item: Adverse Reactions, etc.

Stratification items: Presence or absence of dose change [Absent, present]

for Cabometyx

Breakdown of changes (duplicate [Discontinued (except for

counting) interruption), interrupted, dose

reduced, unknown]

Analytical method: For the above analysis set, frequencies of the number of adverse drug

reactions, etc. will be tabulated for each CTCAE Grade (worst value) of

adverse drug reactions, etc. and stratified by stratification items. Similar

frequency tabulation will be performed for total and CTCAE Grade ≥ 3. For

the incidence of events by stratification factor, the denominator will be the

number of events by CTCAE Grade (worst value). This tabulation will be performed for the overall population and patients treated with Cabometyx

monotherapy and patients treated with nivolumab combination therapy

separately.

### 4.4.3 Administration status of Cabometyx due to adverse events and adverse reactions/infections specified in the safety specifications

### Administration status of Cabometyx due to adverse events included in safety 4.4.3.1 **specifications**

Safety analysis set Analyzed:

Adverse events included in the important identified risks (Hepatic failure, Analysis item:

hepatic function disorder, pancreatitis) in the safety specifications

Presence or absence of dose change Stratification items: [Absent, present]

for Cabometyx

Breakdown of changes (duplicate [Discontinued (except for

counting) interruption), interrupted, dose

reduced, unknown]

Property of Takeda. Analytical method: For the above analysis set, frequencies of the number of adverse events will

be tabulated for each CTCAE Grade (worst value) of adverse events

corresponding to each risk and stratification by the stratification factor.

Similar frequency tabulation will be performed for total and CTCAE Grade ≥

3. For the incidence of events by stratification factor, the denominator will be the number of events by CTCAE Grade (worst value). This tabulation will be

performed for the overall population and patients treated with Cabometyx

monotherapy and patients treated with nivolumab combination therapy

separately.

# 4.4.3.2 Administration status of Cabometyx due to adverse reactions/infections included in safety specifications

Analyzed: Safety analysis set

Analysis item: Adverse reactions, etc. corresponding to important identified risks (Hepatic

failure, hepatic function disorder, pancreatitis) in safety specifications

Stratification items: Presence or absence of dose change [Absent, present]

for Cabometyx

counting) interruption), interrupted, dose

reduced, unknown]

Analytical method: For the above analysis set, frequencies of the number of adverse drug

reactions, etc. will be tabulated for each CTCAE Grade (worst value) of adverse drug reactions, etc. corresponding to each risk and after stratification

by the stratification item. Similar frequency tabulation will be performed for

factor, the denominator will be the number of events by CTCAE Grade (worst

value). This tabulation will be performed for the overall population and patients treated with Cabometyx monotherapy and patients treated with

total and CTCAE Grade  $\geq$  3. For the incidence of events by stratification

nivolumab combination therapy separately.

### 4.5 Factors that may affect safety

# 4.5.1 Status of occurrence of adverse events and adverse drug reactions/infections by patient background and treatment characteristics

Analyzed: Safety analysis set

Analysis item: Adverse Events

Adverse events included in the important identified risks (Hepatic failure,

hepatic function disorder, pancreatitis) in the safety specifications

Adverse Reactions, etc.

Adverse reactions, etc. corresponding to important identified risks (Hepatic

failure, hepatic function disorder, pancreatitis) in safety specifications

Stratification items: Sex [Male, Female]

Age (years) [Min<= - <18, 18<= - <65, 65<= -

<75, 75<= - <85, 85<= - <=Max]

[Min<= - <15, 15<= - <65, 65<= -

<75, 75<= - <85, 85<= - <=Max]

Duration of disease (years)  $[Min \le - <1, 1 \le - \le Max]$ 

Histological diagnosis [Clear cell, non-clear cell, unknown]

| | Clinical Stage | [I, II, III, IV, unknown] |
|---|---|---|
| | (At the start of administration) | |
| | Treatment category | [Outpatient, Inpatient] |
| | (At the start of administration) | |
| | Karnofsky Performance Status Scale | [10<= - <=40, 50<= - <=70, 80<= - |
| | (at the start of treatment) | <=100] |
| | IMDC Risk Categorization | [favorable, intermediate, poor, |
| | (At the start of administration) | unknown] |
| | Metastasis | [Absent, present, unknown] |
| | (At the start of administration) | adlle |
| | Destination of metastasis (multiple | [Brain, lung, liver, bone, lymph node, |
| | counts) | others] |
| | BMI(kg/m2) | [Min<= - <18.5, 18.5<= - <25.0,<br>25.0<= - <30.0, 30.0<= - <=Max] |
| | | 25.0<- <30.0, 30.0<= - <= Max] |
| | History of radiotherapy prior to the | [Absent, present] |
| | start of Cabometyx | <i>J</i> |
| | Anatomical Location (duplicate | [Brain, lung, liver, bone, lymph node, |
| | counting) | others] |
| | Presence/absence of prior systemic | [Absent, present] |
| | drug therapy for renal cell carcinoma | |
| | before the start of Cabometyx (not | |
| | including preoperative or | |
| | postoperative adjuvant drug therapy) | |
| | History of systemic drug therapy for | [Sunitinib, pazopanib, sorafenib, |
| , Tre | renal cell carcinoma before the start of | |
| (0) | Cabometyx (multiple counts) | interferon alpha, nivolumab, |
| 2.05 | | ipilimumab + nivolumab, axitinib + |
| × • | | pembrolizumab, avelumab + axitinib, |
| 800 | | others] |
| | Treatment or surgery for renal cell | [Absent, present] |
| | carcinoma prior to the start of | |
| Property of Takeda. For non-co | Cabometyx | |
| ON THE REAL PROPERTY. | Nephrectomy | [Total nephrectomy, partial |
| 0101 | The status of treatment or surgery for | nephrectomy, no nephrectomy] |
| X | renal cell carcinoma before the start of | |
| | • | |
| | "Present." | |

Presence/absence of history of [Absent, present]
preoperative or postoperative adjuvant
drug therapy before the start of
administration of Cabometyx
When nephrectomy (yes/no) is "total
nephrectomy" or "partial
nephrectomy"

History of preoperative or [Preoperative and postoperative]

postoperative adjuvant drug therapy before the start of administration of Cabometyx (duplicate counting)

Presence or absence of medical [Absent, present]

history

Presence or absence of complications [Absent, present]

Presence or absence of hepatic [Absent, present]

impairment

Presence or absence of renal [Absent, present]

impairment

Cabometyx Starting Dose (mg) [60 mg/day, 40 mg/day, 20 mg/day,

20 mg/day every other day, others]

Analytical method:

Property of Takedai. For non

For the above analysis set, the following analyses should be performed for each stratum of the stratification factor. This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

- (1) Number of subjects with adverse events
- (2) Incidence of adverse events
- (3) Number of patients with adverse events included in the safety specifications
- (4) Incidence of Adverse Events Included in Safety Specifications
- (5) Number of patients with adverse drug reactions, etc.
- (6) Incidence of adverse drug reactions, etc.
- (7) Number of patients with adverse drug reactions, etc. included in safety specifications
- (8) Incidence of adverse drug reactions included in safety specifications
  The following accounting methods will be used for each analysis.
  [Number of patients with adverse events included in adverse events/safety specifications]

• Number of patients with AEs/AEs included in the safety specification. [Incidence of adverse events/adverse events included in safety specifications] It is calculated as the number of patients with adverse events/adverse events included in the safety specification/the number of patients evaluated for safety ×100.

[Number of patients with adverse drug reactions/adverse drug reactions included in the safety specifications]

 Number of patients with adverse drug reactions/adverse drug reactions specified in the safety specification.

[Incidence of adverse drug reactions/adverse drug reactions included in the safety specifications]

Calculate as the number of patients with adverse reactions, etc./adverse reactions, etc. corresponding to the safety specifications/the number of patients evaluated for safety ×100.

### 4.5.2 Incidences of ADRs/infections by gender

Analyzed: Safety analysis set

Analysis item: Adverse Reactions, etc.

Stratification items: Sex [Male, Female]

Analytical method: For the above analytical variable, the analysis of should be performed in the

same manner as in Section 4.1.2 for each of the subgroups of the stratification factors. This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab

combination therapy.

### 4.5.3 Incidences of ADRs and infections by age group

Analyzed: Safety analysis set

Analysis item: Adverse Reactions, etc.

Stratification items: Age [Min<= - <18, 18<= - <65, 65<= -

<75, 75<= - <85, 85<= - <=Max]

[Min<= - <15, 15<= - <65, 65<= -

<75, 75 <= - <85, 85 <= - <= Max

Analytical method: For the above analytical variable, the analysis of should be performed in the

same manner as in Section 4.1.2 for each of the subgroups of the stratification

factors. This tabulation will be performed for the overall population and by

patients receiving Cabometyx monotherapy and patients receiving nivolumab

combination therapy.

### 4.5.4 Status of occurrence of ADRs/infections by presence/absence of hepatic impairment

Safety analysis set Analyzed:

Analysis item: Adverse Reactions, etc.

Stratification items: Presence or absence of hepatic [Absent, present]

impairment

Analytical method: For the above analytical variable, the analysis of should be performed in the

same manner as in Section 4.1.2 for each of the subgroups of the stratification

ins of Use

factors. This tabulation will be performed for the overall population and by patients receiving Cabometyx monotherapy and patients receiving nivolumab

combination therapy.

### 4.5.5 Status of occurrence of ADRs/infections by presence/absence of renal impairment

Analyzed: Safety analysis set

Analysis item: Adverse Reactions, etc.

Stratification items: Presence or absence of renal [Absent, present]

impairment

For the above analytical variable, the analysis of should be performed in the Analytical method:

same manner as in Section 4.1.2 for each of the subgroups of the stratification factors. This tabulation will be performed for the overall population and by Property of Lakeda. For non-commercial patients receiving Cabometyx monotherapy and patients receiving nivolumab

combination therapy.

### **Matters concerning efficacy**

### **Antitumor effect** 5.1

Analyzed: Effectiveness analysis set

Analysis item: Antitumor effect

erms of Use Analytical method: For each of the above analysis items, frequency tabulation of the assessment

results will be performed in the effectiveness analysis set, and the response

rate and 95% confidence interval of the response rate will be calculated. Furthermore, band graphs will be prepared for the above analysis results. This

tabulation is performed separately for patients receiving Cabometyx monotherapy and patients receiving nivolumab combination therapy.

Tumor response by patient background factors and treatment factors

Effectiveness analysis set Analyzed:

Analysis item: Antitumor effect

Stratification items: Sex

Age (years)

Min<= - <18, 18<= - <65, 65<= -

Min<= - <15, 15<= - <65, 65<= -

<75, 75<= - <85, 85<= - <=Max]

Duration of disease (years)  $[Min \le - <1, 1 \le - \le Max]$ 

Histological diagnosis [Clear cell, non-clear cell, unknown]

[I, II, III, IV, unknown]

(At the start of administration)

Karnofsky Performance Status Scale [10<= - <=40, 50<= - <=70, 80<= -

At the start of administ

Karnofsky Performance
(at the start of treatment)

IMDC Risk Categorization
(At the start of administ

Metastasis
(At 1) <=1001

IMDC Risk Categorization [favorable, intermediate, poor,

(At the start of administration) unknown]

[Absent, present, unknown]

(At the start of administration)

Destination of metastasis (multiple [Brain, lung, liver, bone, lymph node,

others]

 $Min \le - <18.5, 18.5 \le - <25.0,$ 

 $25.0 \le -30.0, 30.0 \le -40$ 

History of radiotherapy prior to the [Absent, present]

Presence/absence of prior systemic [Absent, present]

drug therapy for renal cell carcinoma

before the start of Cabometyx (not including preoperative or postoperative adjuvant drug therapy) History of systemic drug therapy for

renal cell carcinoma before the start of Cabometyx (multiple counts)

[Sunitinib, pazopanib, sorafenib, temsirolimus, everolimus, axitinib, interferon alpha, nivolumab,

ipilimumab + nivolumab, axitinib +pembrolizumab, avelumab + axitinib,

others]

Treatment or surgery for renal cell carcinoma prior to the start of

[Absent, present]

Cabometyx

[Total nephrectomy, partial Nephrectomy nephrectomy, no nephrectomy] The status of treatment or surgery for

Cabometyx administration is

renal cell carcinoma before the start of

Presence/absence of history of preoperative or post [Absent, present]

preoperative or postoperative adjuvant drug therapy before the start of administration of Cabometyx

When nephrectomy (yes/no) is "total

[Preoperative and postoperative]

phrectomy (yes
phrectomy" or "partial
nephrectomy"
History of preoperative or
postoperative adjuvant drue
before the start of art
Cabometyx (\*\*
Preser\* postoperative adjuvant drug therapy before the start of administration of Cabometyx (duplicate counting)

Presence or absence of medical [Absent, present]

Presence or absence of complications [Absent, present] Presence or absence of hepatic [Absent, present]

Presence or absence of renal [Absent, present]

Cabometyx [60 mg/day, 40 mg/day, 20 mg/day,

20 mg/day every other day, others]

Analytical method:

Property of Takeda. For non-commercial use only and subject to the applicable Temes of use For each of the above analysis items, frequency tabulation of assessment

35

### Incidences of adverse reactions/infections in the additional pharmacovigilance plan

### Incidences of adverse reactions and infections in the additional pharmacovigilance plan 6.1 (Attached Form 12)

Analyzed: Safety analysis set

ble terms of Use Analysis item: Adverse reactions, etc. included in safety specifications (Important identified risks,

important potential risks, and important missing information)

Stratification Seriousness [Serious, non-serious]

items:

For the above analytical variable, the following analyses should be performed for Analytical

method: each stratum of the stratification factor in accordance with Attached Form 12, (Note)

1~4 of PSEHB/PED Notification No. 0325/10 dated March 25, 2020.

(1) Number of patients with events and incidence

oe in portant iden ation). (a) Takeda. For non-commercial use only and such section of Takeda. Risk names and the order of risk names shall be in accordance with the definitions described in the safety specification (Important identified risks, important potential

### Incidence of adverse reactions/infections in post-marketing surveillance, etc.

### 7.1 Incidence of adverse reactions/infections in post-marketing surveillance, etc. (Attached Form 15)

Analyzed: Safety analysis set

Analysis item: Adverse Reactions, etc.

Analytical For the above analytical variable, the following analyses should be performed.

method:

(1) Status of post-marketing surveillance, etc.

- 1) Number of patients included in safety analysis
- 2) Number of patients with adverse drug reactions, etc.
- Incidence of adverse drug reactions, etc.
- (2) Types of adverse drug reactions, etc.
  - Number of patients with adverse drug reactions, etc. and incidence (by
  - 2) Number of patients with adverse drug reactions, etc. and incidence of them (by PT)

The following accounting methods will be used for each analysis.

[Number of patients with adverse drug reactions, etc.]

Number of patients with adverse drug reactions, etc.

[Incidence of adverse drug reactions, etc.]

Calculate with the number of patients with adverse reactions, etc./the number of patients in the safety analysis set ×100.

[Types of adverse drug reactions, etc.]

- Property of Lakeda: For hon Adverse drug reactions will be coded using MedDRA/J. Data will be broadly classified by SOC, and tabulated by PT within the SOC. If the SOC is "investigations," they will be summarized by HLGT (Sort in ascending order of HLGT code, but not output) and by PT.
  - For SOC, the number of patients with adverse drug reactions, etc. and the incidence should be described in the order of SOC international consensus. A subject who experiences the same SOC more than once will be counted as 1 subject in the SOC.
  - For PT, the number of patients with adverse drug reactions, etc. and the incidence should be entered in ascending order of PT code. If the same PT occurs more than once in the same subject, the subject will be counted as 1 subject in the PT.

\*The "number of patients in the safety analysis set" refers to the "analysis set" (described above) for this analysis.

Propagal of Takeda. For non-commercial use only and subject to the applicable Terms of Use

### Case summary in post-marketing surveillance, etc.

# ect to the applicable Terms of Use 8.1 Case summaries from post-marketing surveillance, etc. (Attached Form 16)

Analyzed: Safety analysis set

Analysis item: Case Number

Name of medical institution

Sex

Age

Reason for use (Disease code and name) Comorbidity (Disease code and name)

Route of Administration

Maximum Dose

Mean dose

Unit

Duration of use (Cabometyx treatment period)

Concomitant medications (Drug code and name)

Degree of efficacy

Reactions (Disease code, name of disease, outcome)

Case Study form No.

Dropout

Reason for Dropout

For the above analytical items, a list will be prepared in accordance with the Analytical

And Attification of the Areda. For non-common of the Areda. guidelines for preparation of reexamination data entry file specified in PSEHB/PED method:

Notification No. 1119 No. 3 dated November 19, 2020.

### **Preparation history (version control)**

| Version | Date | Prepared/changed by | Comments | |
|---|---|---|---|---|
| Original<br>Version | 2024.5.20 | | Preparation of the first version | ~ |

Properly of Takeda, For non-commercial use only and subject to the applicable Terms of Use

[Appendix 1] Comparison Table of Changes

| | | After amendment Reason for change | | |
|---|---|---|---|---|
| Page | Before change | After amendment | 2061 | Reason for change |
| | | | 10. | |
| | | | H | |
| | | | , | |
| | | 4 5 1/4 | | |
| | | and | | |
| | | lh. | | |
| | | , use | | |
| | | cial | | |
| | | ele | | |
| | Olul, | | | |
| | 7.00 | | | |
| | 100 | | | |
| | <b>₹</b> 0′ | | | |
| | ×ò·` | | | |
| | of solutions and solutions are solutions and solutions are solutions and solutions are solutions are solutions. | | | |
| | × 10. | | | |
| | "1°", | 1 | | |
| | 5(,) | | | |
| orok | Before change Before change Before change Before change | | | |
| X | | | | |